CLINICAL TRIAL: NCT01419262
Title: DO IT Trial: Vitamin D Outcomes and Interventions In Toddlers
Acronym: DO IT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Mount Sinai Hospital, Canada (Other); Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Jonathon L Maguire, Physician/ Principal Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1000025147
Record Dates: First submitted 2011-08-16; First posted 2011-08-18 (Estimated); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Respiratory Tract Infections; Asthma; Avitaminosis
Keywords: Vitamin D; Randomized Controlled Trial; Child, Preschool; Dietary Supplements; Respiratory Tract Infections; Asthma
MeSH Terms: conditions — Respiratory Tract Infections; Asthma; Avitaminosis | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2000 IU per day vitamin D (Experimental)
  Interventions: Drug: Vitamin D3 - Cholecalciferol 2000 IU
- 400 IU per day vitamin D (Active Comparator)
  Interventions: Drug: Vitamin D - Cholecalciferol 400 IU

INTERVENTIONS:
Drug: Vitamin D - Cholecalciferol 400 IU — One drop per day (liquid), 400 IU, 4 to 9 months depending on date of enrollment and date of follow-up
  Other Names: Baby Ddrops; Health Canada NPN #80001869
  Arms: 400 IU per day vitamin D
Drug: Vitamin D3 - Cholecalciferol 2000 IU — One drop per day (liquid), 2000 IU, 4 to 9 months depending on date of enrollment and date of follow-up
  Other Names: Ddrops 2000 IU
  Arms: 2000 IU per day vitamin D

SUMMARY:
Vitamin D can be made in the skin by exposure to sunlight and can be found in certain foods. Vitamin D levels are alarmingly low in many North American children. Several health issues have been linked with low vitamin D. These include colds caused by viruses and asthma attacks. However, no study has determined whether vitamin D supplementation can reduce the risk of these conditions in young children where they are most common and most severe.

The goals of this study are to determine whether wintertime high dose vitamin D supplementation of preschoolers can prevent colds and asthma attacks. The investigators also aim to work out how much money would be saved by the health care system and society if preschoolers were routinely supplemented with Vitamin D during the winter. The investigators believe that preschoolers receiving 'high dose' vitamin D supplementation during the wintertime will be less likely to have colds, asthma attacks, and low vitamin D levels and will be less likely to use the medical system and keep their parents away from work.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy children by parental report
2. Have reached their 1st birthday but not past their 6th birthday
3. Present to a TARGet Kids! practice for routine primary healthcare prior to viral season (September through November)
4. Parents provide informed consent to participate.

Exclusion Criteria:

1. Children with gestational age < 32 weeks
2. Children with chronic illness (except for asthma) on parental report which is known to interfere with vitamin D metabolism and increase the risk of respiratory infection
3. Children with a sibling participating in the study to reduce clustering effects.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 703 (Actual)
Dates: Start 2011-09; Primary Completion 2015-05 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Number of Laboratory confirmed upper respiratory tract infections | Up to 8 months
  Parents of enrolled children will be asked to obtain a nasal swab from their child and complete a symptom checklist with each URTI. Reverse transcriptase polymerase chain reaction will be performed on each sample. Samples will be tested for 18 common respiratory viruses using the ID-TagTM RVP assay using the Luminex xMAPTM system.

SECONDARY OUTCOMES:
Number of parent reported upper respiratory tract infections | Up to 8 months
  Parental reported URTI symptoms will be defined as two or more of fever, cough, runny nose, sore throat, headache, vomiting, feels unwell, muscle aches, ear ache or infection, poor appetite, not sleeping well, cranky/fussy, low energy or crying more than usual from a validated parent completed symptom checklist.
Number of Asthma exacerbations | Up to 8 months
  Asthma exacerbation will be defined as a wheezing episode in children with asthma as obtained from parent completed symptom checklist based on the International Study of Asthma and Allergies in Childhood (ISAAC).
Serum vitamin D level | 5-8months
  Blood for serum levels will be drawn by trained pediatric phlebotomists from for determination of 25-hydroxyvitamin D. Total 25-hydroxyvitamin D will be measured from serum samples using a competitive two-step chemiluminescence assay.
Direct and indirect economic costs associated with upper respiratory tract infections | 16 months
  Cost-consequence and cost-effectiveness analyses will be conducted using data from this clinical trial. A societal perspective will be employed as both direct health service utilization costs as well as indirect costs to families from URTI will be calculated for the 400 IU per day versus 2000 IU per day groups.

OTHER OUTCOMES:
Body Mass index z-score | Up to 8 months
  Weight and height will be measured at both study baseline and follow-up by trained research assistants. BMI will be determined by dividing the children's measured weight (kg) by height (m2). The BMI z-score [zBMI] will be determined using the World Health Organization Growth standards, standardized for age and sex.
Waist circumference z-score | Up to 8 months
  Waist circumference will be measured at both study baseline and follow-up by trained research assistants. Waist circumference will be measured at the mid-axillary line above the right iliac crest. Waist circumference z-score will be calculated internally within the entire TARGet Kids! study cohort.
Serum Lipids | Up to 8 months
  Blood for serum levels will be drawn by trained pediatric phlebotomists from for determination of total cholesterol, low-density lipoprotein [LDL] cholesterol, high-density lipoprotein [HDL] cholesterol and non-HDL cholesterol.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathon L Maguire, MD, MSc, Principal Investigator — St. Michael's Hospital, Toronto, Ontario, Canada
Locations (2):
- Canada (2):
  - St. Michael's Hospital, Toronto, Ontario
  - Hospital for Sick Children, Toronto, Ontario

REFERENCES:
- [Derived] Huey SL, Acharya N, Silver A, Sheni R, Yu EA, Pena-Rosas JP, Mehta S. Effects of oral vitamin D supplementation on linear growth and other health outcomes among children under five years of age. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD012875. doi: 10.1002/14651858.CD012875.pub2. PMID 33305842
- [Derived] Aglipay M, Birken CS, Parkin PC, Loeb MB, Thorpe K, Chen Y, Laupacis A, Mamdani M, Macarthur C, Hoch JS, Mazzulli T, Maguire JL; TARGet Kids! Collaboration. Effect of High-Dose vs Standard-Dose Wintertime Vitamin D Supplementation on Viral Upper Respiratory Tract Infections in Young Healthy Children. JAMA. 2017 Jul 18;318(3):245-254. doi: 10.1001/jama.2017.8708. PMID 28719693